CLINICAL TRIAL: NCT04025021
Title: Targeted Fortification of Human Breast Milk and Adjustment of TPN for Very Low Birth Weight Infants to Optimize Growth and Nutrition Using the Miris Mid-infrared Human Milk Analyzer
Brief Title: Targeted Breast Milk Fortification for Very Low Birth Weight Infants in the NICU
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to enroll patients, sample collection
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Sharon Groh-Wargo, Principal Investigator, Neonatal Nutritionist, Clinical Professor, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-00200
Record Dates: First submitted 2019-07-10; First posted 2019-07-18 (Actual); Results first posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-01

CONDITIONS: Human Milk; Neonate; Breast Milk
Keywords: Targeted Fortification; Human Milk Analysis; Neonatal Nutrition

STUDY DESIGN:
Intervention Model Description: This study will be a randomized control trial with 2 arms: control group (standard fortification) or intervention group (targeted fortification) in a 1:1 allocation ratio. Allocation group will be stratified to four groups according to birth weight: <750g, 751-1000g, 1001-1250g, 1251-1500g. This stratification is based upon our NICU feeding guideline, and will ensure that enrolled infants will receive comparable nutrition progression (e.g. NPO (nil per os) days, days of trophic feeds) throughout the study period. The allocation will be concealed in a sequentially numbered, opaque, sealed envelope, that will be opened after consent is obtained.
Masking Description: After randomization, the groups will not be blinded to the investigators or caregivers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control group (standard fortification) (No Intervention): Breast milk will be fortified standard with Similac Human Milk Fortifier 1 packet:
  50 ml breast milk at 50ml/kg/day enteral feeds, then 1 packet:25 ml breast milk at 75 ml/kg/day. As feedings are advanced to goal of 150 ml/kg/day, the TPN and SMOF lipids (Fat Emulsion Comprised of Soy Oil, Medium Chain Triglycerides, Olive Oil, and Fish Oil) will be decreased per standard management and NICU guidelines.
- Intervention group (targeted fortification) (Experimental): Breast milk will be fortified standard with Similac Human Milk Fortifier 1 packet:
  50 ml breast milk at 50ml/kg/day enteral feeds, then 1 packet:25 ml breast milk at 75 ml/kg/day. During this time, as the volume decreases, the TPN and SMOF lipids will be optimized to provide a goal of 4 g/kg/day of protein, and 100-130kcal/kg/day. At 100 ml/kg/day of enteral feeds additional liquid protein and/or microlipids will be added to the breast milk to provide goal of 4 g/kg/day of protein and 100-130 kcal/kg/day. This will be determined by analysis of the milk and reported composition. They will continue targeted fortification for 4 weeks after achieving full feeds of 150 ml/kg/day. Breast milk analysis will occur on a weekly basis immediately after birth for all infants enrolled in the study.
  Interventions: Dietary Supplement: Targeted Fortification; Device: The Miris Human Milk Analyzer

INTERVENTIONS:
Dietary Supplement: Targeted Fortification — The TPN and SMOF lipids will be optimized to provide a goal of 4 g/kg/day of protein, and 100-130kcal/kg/day. At 100 ml/kg/day of enteral feeds additional liquid protein and/or microlipids will be added to the breast milk to provide goal of 4 g/kg/day of protein and 100-130 kcal/kg/day. This will be determined by analysis of the milk and reported composition. They will continue targeted fortification for 4 weeks after achieving full feeds of 150 ml/kg/day.
  Arms: Intervention group (targeted fortification)
Device: The Miris Human Milk Analyzer — The Miris human milk analyzer is a mid infrared that reports the amount of energy absorbed at each wavelength. The amount of fat (grams), lactose (grams), total protein (grams), true protein (grams), and energy (kcal) per 100 ml will be reported.
  Arms: Intervention group (targeted fortification)

SUMMARY:
This study evaluates the effectiveness of individualized human milk fortification for very low birth weight (<1500 g) babies in the NICU (Neonatal Intensive Care Unit) to optimize their growth. Breast milk analysis will occur on a weekly basis using the Miris Human Milk Analyzer. In the Control group, participants will receive standard TPN (total parenteral nutrition) and lipids and breast milk fortification according to MetroHealth's NICU guidelines. The Intervention group will receive TPN and lipids optimized depending on the results of breast milk analysis, followed by additional individualized fortification using additional microlipids and/or liquid protein to achieve the goal of 4g protein/kg/day and 100-130 kcal/kg/day.

DETAILED DESCRIPTION:
Human milk has a variety of benefits for neonates, especially premature neonates, including a decreased risk of for necrotizing enterocolitis, sudden infant death syndrome (SIDS), respiratory syncytial virus (RSV) bronchiolitis, respiratory infections, and many other childhood conditions. There is variability in macronutrient and caloric content of breast milk between mothers, making it difficult to accurately quantify the nutritional content the breast milk is providing. The protein content varies by postnatal age, and the fat content varies temporally during a feed. Currently calculations use a standard value for caloric density and macronutrient content of breast milk, which is a reported average, but not necessarily specific to each individual mother. Human milk analysis has been used to address this variability. The Miris Human Milk Analyzer (HMA) is a mid-infrared analyzer and has been evaluated in many studies. It measures the macronutrient content of breast milk, providing values for protein, fat, carbohydrates, and calculated calories. By having this information available, the fortification added to breast milk can be tailored specifically to each mother's breast milk composition to meet each neonate's nutritional needs, and optimize growth.This will be a prospective randomized control study of preterm infants less than 1500 grams [very low birth weight (VLBW)] receiving human milk (maternal or donor) will be included. The control group will receive adjustment of total parenteral nutrition (TPN) per NICU guidelines as enteral feedings are advanced followed by standard fortification of human milk. The intervention group will have TPN (protein and lipids) adjusted based on analysis of human milk as feedings are advanced to provide goal 4g/kg/day of protein and 100-130 kcal/kg/day followed by targeted fortification of breast milk based on human milk analysis to continue to provide 4 g/kg/day of protein and 100-130 kcal/kg/day for once full feeds are achieved. The primary aim of this study is to evaluate the growth, anthropometric measurements, and body composition, to see if targeted fortification improves neonatal growth. By optimizing neonatal growth and nutrition there is potential to also have an impact on other morbidities and long term neurodevelopmental outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Premature infants <1500 g
* Mother consenting to provide breast milk or use of donor breast milk

Exclusion Criteria:

* Infants with major congenital malformations
* Infants with medical conditions precluding them from having breast milk
* Mothers with medical conditions that preclude them form providing breast milk
* Insufficient breast milk supply
* Refusal of donor breast milk
* Mother is non-English speaking

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Groh-Wargo, PhD, RDN, Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Section on Breastfeeding. Breastfeeding and the use of human milk. Pediatrics. 2012 Mar;129(3):e827-41. doi: 10.1542/peds.2011-3552. Epub 2012 Feb 27. PMID 22371471
- [Background] Martin CR, Ling PR, Blackburn GL. Review of Infant Feeding: Key Features of Breast Milk and Infant Formula. Nutrients. 2016 May 11;8(5):279. doi: 10.3390/nu8050279. PMID 27187450
- [Background] Fusch G, Kwan C, Kotrri G, Fusch C. "Bed Side" Human Milk Analysis in the Neonatal Intensive Care Unit: A Systematic Review. Clin Perinatol. 2017 Mar;44(1):209-267. doi: 10.1016/j.clp.2016.11.001. Epub 2016 Dec 29. PMID 28159207
- [Background] Tudehope DI. Human milk and the nutritional needs of preterm infants. J Pediatr. 2013 Mar;162(3 Suppl):S17-25. doi: 10.1016/j.jpeds.2012.11.049. PMID 23445843
- See also: Miris HMA, Human Milk Analyzer website — http://mirissolutions.com/solution

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group (Targeted Fortification): Breast milk (BM) will be fortified standard with Similac Human Milk Fortifier 1 packet:
  50 ml BM at 50ml/kg/day enteral feeds, then 1 packet:25 ml breast milk at 75 ml/kg/day. During this time, as the volume decreases, the TPN and SMOF lipids will be optimized to provide a goal of 4 g/kg/day of protein, and 100-130kcal/kg/day. At 100 ml/kg/day of enteral feeds additional liquid protein and/or lipids will be added to the breast milk to provide goal of 4 g/kg/day of protein and 100-130 kcal/kg/day. This will be determined by analysis of the milk and reported composition. They will continue targeted fortification for 4 weeks after achieving full feeds of 150 ml/kg/day. BM analysis will occur on a weekly basis immediately after birth for all infants enrolled in the study.
  Targeted Fortification: parenteral nutrition will be optimized to provide a goal of 4 g/kg/day of protein, and 100-130kcal/kg/day. At 100 ml/kg/day of enteral feeds additional protein and/or fat will be added to the breast milk to provide goal of 4 g/kg/day of protein and 100-130 kcal/kg/day. This will be determined by analysis of the milk and reported composition. They will continue targeted fortification for 4 weeks after achieving full feeds of 150 ml/kg/day.
Period: Overall Study
Arm/Group | Control Group (Standard Fortification) | Intervention Group (Targeted Fortification)
Started | 2 | 1
Completed | 0 | 0
Not Completed | 2 | 1
Not completed — Study discontinued with onset of COVID-19 pandemic | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Intervention Group (Targeted Fortification): Breast milk will be fortified standard with Similac Human Milk Fortifier 1 packet:
  50 ml breast milk at 50ml/kg/day enteral feeds, then 1 packet:25 ml breast milk at 75 ml/kg/day. During this time, as the volume decreases, the TPN and SMOF lipids will be optimized to provide a goal of 4 g/kg/day of protein, and 100-130kcal/kg/day. At 100 ml/kg/day of enteral feeds additional liquid protein and/or microlipids will be added to the breast milk to provide goal of 4 g/kg/day of protein and 100-130 kcal/kg/day. This will be determined by analysis of the milk and reported composition. They will continue targeted fortification for 4 weeks after achieving full feeds of 150 ml/kg/day. Breast milk analysis will occur on a weekly basis immediately after birth for all infants enrolled in the study.
  Targeted Fortification: The TPN and SMOF lipids will be optimized to provide a goal of 4 g/kg/day of protein, and 100-130kcal/kg/day. At 100 ml/kg/day of enteral feeds additional liquid protein and/or microlipids will be added to the breast milk to provide goal of 4 g/kg/day of protein and 100-130 kcal/kg/day. This will be determined by analysis of the milk and reported composition. They will continue targeted fortification for 4 weeks after achieving full feeds of 150 ml/kg/day.
- Total: Total of all reporting groups
Arm/Group | Control Group (Standard Fortification) | Intervention Group (Targeted Fortification) | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Continuous [Mean (Full Range); unit: weeks] | 28.5 [25 to 32.4] | 29 [29 to 29] | 28.8 [25 to 32.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 0 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Body Composition
Description: Body composition will be measured by air displacement plethysmography (PEAPod). As standardized assessment of body composition is relatively new in the preterm infant population, we are using clinical judgment to determine that a difference in fat free mass z-score (from data from Norris T, 2019) of 0.5 is clinically significant.
Time Frame: 4 weeks after baby reaches full feeds (150 mL/kg/day) or at NICU discharge
Population: Study discontinued due to onset of COVID pandemic. No data were collected for this Outcome Measure.
Arm/Group | Control Group (Standard Fortification) | Intervention Group (Targeted Fortification)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Weight Gain Velocity
Description: Weight gain velocity, measured in grams/kg/day
Time Frame: From enrollment in study to 4 weeks after full feeds (150 mL/kg/day) or at NICU discharge.
Population: Study discontinued due to onset of COVID pandemic. No data were collected for this Outcome Measure.
Arm/Group | Control Group (Standard Fortification) | Intervention Group (Targeted Fortification)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Weight Gain
Description: Daily weight will be obtained, measured in grams
Time Frame: From enrollment in study to 4 weeks at full feeds (150 mL/kg/day) or at NICU discharge.
Population: Study discontinued due to onset of COVID pandemic. No data were collected for this Outcome Measure.
Arm/Group | Control Group (Standard Fortification) | Intervention Group (Targeted Fortification)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Linear Growth
Description: Weekly measurements of length will be obtained throughout the study, measured in centimeters
Time Frame: From enrollment in study to 4 weeks at full feeds (150 mL/kg/day) or at NICU discharge.
Population: Study discontinued due to onset of COVID pandemic. No data were collected for this Outcome Measure.
Arm/Group | Control Group (Standard Fortification) | Intervention Group (Targeted Fortification)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Head Circumference Growth
Description: Weekly measurements of head circumference will be obtained throughout the study, measured in centimeters
Time Frame: From enrollment in study to 4 weeks at full feeds (150 mL/kg/day) or at NICU discharge.
Population: Study discontinued due to onset of COVID pandemic. No data were collected this Outcome Measure.
Arm/Group | Control Group (Standard Fortification) | Intervention Group (Targeted Fortification)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Body Composition
Description: Mid upper arm circumference (cm) or skinfold thickness (mm) will be measured weekly throughout the study and combined with length to calculate the body composition
Time Frame: From enrollment in study to 4 weeks at full feeds (150 mL/kg/day) or at NICU discharge.
Population: Study discontinued due to onset of COVID pandemic. No data were collected for this Outcome Measure.
Arm/Group | Control Group (Standard Fortification) | Intervention Group (Targeted Fortification)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 0 days
Description: Study discontinued due to onset of COVID pandemic. No data were collected for Adverse Events.
Arm/Group | Control Group (Standard Fortification) | Intervention Group (Targeted Fortification)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Early termination of the study due to the onset of the COVID pandemic. As a result, no data were analyzed or collected from participants enrolled. Therefore, there are no data to provide for outcome measures and adverse events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-19): https://cdn.clinicaltrials.gov/large-docs/21/NCT04025021/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/21/NCT04025021/ICF_001.pdf